CLINICAL TRIAL: NCT03885050
Title: Modified Ross Score for Evaluation of Heart Failure in Children With Lower Respiratory Tract
Brief Title: Modified Ross Score for Evaluation of Heart Failure in Children
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Enas Saad Hassan, Principal investigator, Assiut University
Other Study IDs: MRS
Record Dates: First submitted 2019-03-16; First posted 2019-03-21 (Actual); Last update posted 2019-03-21 (Actual); Status verified 2019-03

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Ross score — modified score used for evaluation of heart failure in children, as a diagnostic tool for severity of heart failure

SUMMARY:
* Identification of Patient those at risk For heart failure associated with lower respiratory tract infection
* Assess the value of Ross score evaluation in lower respiratory tract infection complicated with HF, as a diagnostic tool for severity of HF

DETAILED DESCRIPTION:
- Pneumonia in young children remains a global epidemic and a leading cause of death in under-5 children. The annual incidence is approximately 156 million patients worldwide; and pneumonia and its complications led to approximately 0.92 million under-5 deaths in 2015.

In adult patients, cardiac events such as congestive heart failure (CHF) are among the leading complications associated with increased morbidity and mortality, but the association in pediatric patients is not well Established

At Suratthani Hospital, Thailand study therefore investigated the characteristics and factors associated with CHF in under-5 children with pneumonia and respiratory failure (RF). Also, revealed that Pneumonia with respiratory failure is associated with CHF even in healthy children without cardiac risks. The awareness and early recognition of CHF, particularly in male, and bacterial pneumonia is important in order to provide immediate treatment to reduce complications.

- A diagnosis of heart failure due to right ventricular affection requires a high index of suspicion since symptoms of heart failure such as easy fatiguability and tachypnoea are obscured by the primary pulmonary disease itself.6 The American Heart Association recommends early echocardiographic studies to diagnose pulmonary hypertension in children with obstructive apnea and sickle cell anaemia.2 Systolic pulmonary artery pressure can be estimated by echocardiographic Doppler assessment using definition of mean pulmonary artery pressure of >25mmHg. A ten-year review of chronic cor pulmonale secondary to respiratory diseases in Ghana was propelled by the fact that early diagnosis can lead to treatment of the respiratory disease, which would then improve a child's cardiac status. Nine cases of chronic cor pulmonale secondary to respiratory diseases were admitted during the period. Three had bronchiectasis as shown in Table 1. Of the three with bronchiectasis, one had congenital lung aplasia; one had a repair of tracheoesophageal atresia at the age of one week. The other was HIV-positive with bronchiectasis secondary to pulmonary tuberculosis.

Children with right heart failure should be investigated for pulmonary cause since early recognition and treatment would improve outcome

Until 1987, the only system available for grading HF in children was the New York Heart Association (NYHA) classification. However, this system was based on limitations to physical activity for adults, which did not translate well for use with children, particularly infants.2 Therefore, we developed a symptom-based classification using more age-appropriate variables. new Ross HF classification from grades I to IV

Several authors have modified Ross scoring system to expand its use to older children.

with all this recent data on factors predictive of outcomes in children with HF that a revision in how we grade symptom severity is required. It also is apparent that age stratification is required to encompass the changes in signs and symptoms that children manifest from infancy to late childhood. A classification system should include the biomarkers, echo parameters of systolic function and mitral or systemic atrioventricular valve (AV) insufficiency, and reflect exercise limitations reflected by feeding and growth in infants and exercise capacity indicated by percentage of predicted maximal oxygen uptake (VO2) in older children. Therefore an age-based Ross classification using the original variables that proved to be sensitive and specific and adding the new evidence-based data.

ELIGIBILITY:
Inclusion Criteria:

* Children with respiratory lower tract infection

Exclusion Criteria:

* Patients with past history of cardiac disease
* Patients with past history of renal disease.
* Patient less than 1 month
* Parent refusal to participate the research

Ages: 1 Month to 18 Years | Sex: All
Age Groups: Child, Adult
Study Population: Infants and children around age of (1month to 18 years old) admitted in the Intensive Care Unit and Intermediate Care Unit in Assiut Pediatric Hospital in a period of 6 months
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2019-11-01 (Estimated); Primary Completion 2020-05-30 (Estimated); Study Completion 2020-09-30 (Estimated)

PRIMARY OUTCOMES:
The mean score in the study population | 1 hour
  Modified Ross Score For Evaluation of Heart Failure in Children with Lower Respiratory Tract Infection Admitted To Assiut University Pediatric Hospital

REFERENCES:
- [Background] Laer S, Mir TS, Behn F, Eiselt M, Scholz H, Venzke A, Meibohm B, Weil J. Carvedilol therapy in pediatric patients with congestive heart failure: a study investigating clinical and pharmacokinetic parameters. Am Heart J. 2002 May;143(5):916-22. doi: 10.1067/mhj.2002.121265. PMID 12040358
- [Background] Ross RD. The Ross classification for heart failure in children after 25 years: a review and an age-stratified revision. Pediatr Cardiol. 2012 Dec;33(8):1295-300. doi: 10.1007/s00246-012-0306-8. Epub 2012 Apr 5. PMID 22476605
- [Background] Ross RD, Bollinger RO, Pinsky WW. Grading the severity of congestive heart failure in infants. Pediatr Cardiol. 1992 Apr;13(2):72-5. doi: 10.1007/BF00798207. PMID 1614922
- [Background] Corrales-Medina VF, Musher DM, Wells GA, Chirinos JA, Chen L, Fine MJ. Cardiac complications in patients with community-acquired pneumonia: incidence, timing, risk factors, and association with short-term mortality. Circulation. 2012 Feb 14;125(6):773-81. doi: 10.1161/CIRCULATIONAHA.111.040766. Epub 2012 Jan 4. PMID 22219349
- [Background] Musher DM, Rueda AM, Kaka AS, Mapara SM. The association between pneumococcal pneumonia and acute cardiac events. Clin Infect Dis. 2007 Jul 15;45(2):158-65. doi: 10.1086/518849. Epub 2007 Jun 6. PMID 17578773